CLINICAL TRIAL: NCT02111785
Title: The DECS Trial: DExamethasone Versus Burr Hole Craniostomy for Symptomatic Chronic Subdural Hematoma
Brief Title: Dexamethasone Versus Burr Hole Craniostomy for Symptomatic Chronic Subdural Hematoma
Acronym: DECS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Accrual too slow; Study P.I. passed away.
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17294
Record Dates: First submitted 2014-04-03; First posted 2014-04-11 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Chronic Subdural Hematoma
Keywords: Dexamethasone; Burr hole craniostomy; Chronic subdural hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Burr Hole Craniostomy randomized (Active Comparator): Group receiving burr hole craniostomy and drainage of chronic subdural hematoma
  Interventions: Procedure: Burr Hole Craniostomy
- Dexamethasone randomized (Experimental): Dexamethasone, tablet, initial dose 4mg q8h, total duration 15 days
  Interventions: Drug: Dexamethasone
- Burr hole craniostomy observational (Other): Observational cohort of patients selecting burr hole craniostomy
  Interventions: Procedure: Burr Hole Craniostomy
- Dexamethasone observational (Other): Observational cohort of patients treated with dexamethasone protocol
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Treatment with a short course of oral dexamethasone
  Other Names: dex
  Arms: Dexamethasone observational; Dexamethasone randomized
Procedure: Burr Hole Craniostomy — Treatment with surgical burr hole craniostomy and evacuation of SDH
  Other Names: Burr hole drainage
  Arms: Burr Hole Craniostomy randomized; Burr hole craniostomy observational

SUMMARY:
Chronic subdural hematoma (cSDH) is condition where blood has slowly leaked out of small blood vessels surrounding the brain. Over time, the blood may cause a variety of symptoms including headache, confusion, limb weakness, and difficulty speaking.

There is currently no agreement among physicians as to the best way to treat this condition.

The study hypothesis to be tested was: For patients with unilateral, symptomatic chronic subdural hematoma, there is no difference in clinical outcomes, as measured by achievement of modified Rankin Score of 0-2 at 6 months, between those treated with a 2 week course of oral dexamethasone, compared with those treated with burr hole surgical drainage.

DETAILED DESCRIPTION:
Chronic subdural hematoma (cSDH) is condition where blood has slowly leaked out of small blood vessels surrounding the brain. Over time, the blood may cause a variety of symptoms including headache, confusion, limb weakness, and difficulty speaking.

There is currently no agreement among physicians as to the best way to treat this condition. One option is to do a surgery to drain the blood that has collected. Usually the surgery involves drilling small holes in the skull to relieve pressure and allow blood and fluids to be drained. Another option is to give medications such as steroids that might reduce the swelling. However, no drugs have been approved by the Food and Drug Administration (FDA) specifically to treat this condition. Some patients elect to have no treatment.

The purpose of this study was to investigate whether investigational treatment with a 2 week course of oral dexamethasone is as effective as surgery for cSDH. The study hypothesis to be tested was: For patients with unilateral, symptomatic chronic subdural hematoma, there is no difference in clinical outcomes, as measured by achievement of modified Rankin Score of 0-2 at 6 months, between those treated with a 2 week course of oral dexamethasone, compared with those treated with burr hole surgical drainage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18 years of age or older
* Informed consent obtained from a patient or a legal representative before enrollment
* Enrollment into the study within 12 hours of detection of chronic subdural hematoma on cranial imaging
* Presence of symptoms referable to chronic subdural hematoma, including one or more of the following: Headache; altered mental status, limb weakness, dysphasia, or focal neurological deficit
* Demonstration of unilateral chronic subdural hematoma on cranial imaging, including the following features: On computed tomography imaging, iso- or hypo-intensity extra-axial collection with or without presence of acute component; radiologic interpretation of magnetic resonance imaging consistent with subacute or chronic SDH; with or without evidence of acute hemorrhagic component
* Maximum depth of subdural hematoma of less than 20mm, with less than 10mm of midline shift, as measured on axial CT or MR imaging
* Absence of skull fracture over the subdural hematoma
* Able to receive the drug treatment

Exclusion Criteria:

* Presence of skull fracture over the subdural hematoma, or other specific etiology for cSDH not suitable for drainage by burr hole craniostomy, such as presence of a ventriculoperitoneal shunt
* Extent of subdural hematoma > 20mm in maximal depth, or > 10mm of midline shift, as measured on axial CT or MR imaging
* GCS <8 or cSDH of an extent or size for which craniotomy, rather than burr hole drainage alone, is judged necessary by the neurosurgery attending on call
* Prior diagnosis of dementia
* Presence of symptomatic peptic ulcer, psychosis, active or suspected TB, acute infection, or documented hypersensitivity or allergy to dexamethasone
* Pregnancy (confirmed by a serum human chorionic gonadotropin pregnancy test) or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer De Jong, Study Director — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Burr Hole Craniostomy Randomized: Group receiving burr hole craniostomy and drainage of chronic subdural hematoma
  Burr Hole Craniostomy
- Dexamethasone Randomized: Dexamethasone, tablet, initial dose 4mg q8h, total duration 15 days
  Dexamethasone
- Burr Hole Craniostomy Observational: Observational cohort of patients selecting burr hole craniostomy
  Burr Hole Craniostomy
- Dexamethasone Observational: Observational cohort of patients treated with dexamethasone protocol
  Dexamethasone
Period: Overall Study
Arm/Group | Burr Hole Craniostomy Randomized | Dexamethasone Randomized | Burr Hole Craniostomy Observational | Dexamethasone Observational
Started | 3 | 5 | 1 | 1
Completed | 3 | 4 | 1 | 1
Not Completed | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population represents patients meeting inclusion/exclusion criteria who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Burr Hole Craniostomy Randomized | Dexamethasone Randomized | Burr Hole Craniostomy Observational | Dexamethasone Observational | Total
Number analyzed (Participants) | 3 | 5 | 1 | 1 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 0 | 0 | 3
  >=65 years | 1 | 4 | 1 | 1 | 7
Age, Continuous [Mean (Full Range); unit: years] | 75.3 [54 to 88] | 72.6 [47 to 87] | 76 [76 to 76] | 74 [74 to 74] | 73.3 [47 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 5 | 1 | 1 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 1 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Modified Rankin Score of 0, 1 or 2
Description: The Modified Rankin Scale (mRS)
  The mRS is evaluated as follows:
  0 - No symptoms
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
  Higher scores on the mRS scale mean a worse outcome.
Time Frame: 6 months after diagnosis
Population: Number of Participants with a modified Rankin Score of 0, 1 or 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Burr Hole Craniostomy Randomized | Dexamethasone Randomized | Burr Hole Craniostomy Observational | Dexamethasone Observational
Number analyzed (Participants) | 3 | 5 | 1 | 1
Participants | 3 | 4 | 1 | 1

2. Secondary Outcome: Rate of Treatment Failure
Description: This measure includes rate of repeat surgery in the burr hole group and rate of progression to surgery in the dexamethasone group
Time Frame: 6 months after diagnosis
Population: Reflects population analyzed for treatment failure. The one patient in the dexamethasone randomized group who died was not analyzed for this secondary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Burr Hole Craniostomy Randomized | Dexamethasone Randomized | Burr Hole Craniostomy Observational | Dexamethasone Observational
Number analyzed (Participants) | 3 | 4 | 1 | 1
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Participants With Modified Rankin Score 0, 1 or 2 at 6 Months
Description: as for outcome 1
Time Frame: 6 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Burr Hole Craniostomy Randomized | Dexamethasone Randomized | Burr Hole Craniostomy Observational | Dexamethasone Observational
Number analyzed (Participants) | 3 | 5 | 1 | 1
Participants | 3 | 4 | 1 | 1

4. Secondary Outcome: Participants With a Glasgow Coma Scale Score of 15 at 6 Month Follow-up
Description: Glasgow Coma Scale (GCS) The GCS is evaluated on a scale from 3 to 15, with higher scores indicating better outcome.
Time Frame: 6 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Burr Hole Craniostomy Randomized | Dexamethasone Randomized | Burr Hole Craniostomy Observational | Dexamethasone Observational
Number analyzed (Participants) | 3 | 5 | 1 | 1
Participants | 3 | 4 | 1 | 1

5. Secondary Outcome: Participants With a Markwalder Grading Score of 0
Description: Markwalder Grading Score (MGS)
  The MGS is assessed as follows:
  Grade 0 - Patient neurologically normal Grade 1 - Patient alert and oriented; mild symptoms, such as headache; absent or mild symptoms or neurologic deficit, such as reflex asymmetry Grade 2 - Patient drowsy or disoriented with variable neurological deficit, such as hemiparesis Grade 3 - Patient stuporous but responding appropriately to noxious stimuli; several focal signs, such as hemiparesis Grade 4 - Patient comatose with absent motor response to painful stimuli; decerebrate or decorticate posturing.
  Higher scores mean a worse outcome.
Time Frame: 6 months after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Burr Hole Craniostomy Randomized | Dexamethasone Randomized | Burr Hole Craniostomy Observational | Dexamethasone Observational
Number analyzed (Participants) | 3 | 5 | 1 | 1
Participants | 3 | 4 | 1 | 1

6. Other Pre Specified Outcome: Rate of Radiographic Resolution of Chronic Subdural Hematoma
Description: The data were not collected.
Time Frame: 6 months after diagnosis
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events assessed included number of participants experiencing infection, seizure, medication intolerance, DVT and PE.
Arm/Group | Burr Hole Craniostomy Randomized | Dexamethasone Randomized | Burr Hole Craniostomy Observational | Dexamethasone Observational
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/5 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT02111785/Prot_SAP_000.pdf